CLINICAL TRIAL: NCT05967182
Title: A Single-Arm Study of Pembrolizumab With Gemcitabine and Cisplatin as Perioperative Therapy for Potentially Resectable Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1003; NCI-2023-05889 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — pembrolizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab with Gemcitabine and Cisplatin (Experimental): Participants will receive 4 cycles (21 days each) of the combined chemotherapy before and after your scheduled surgery. During the 9 months of chemotherapy treatment, participants will have clinic visits every 3 weeks or so. During the 2-4 year follow-up period, participants will come to the clinic every 3 months or so
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Pembrolizumab — Given by IV (vein)
Drug: Gemcitabine — Given by IV (vein)
Drug: Cisplatin — Given by IV (vein)

SUMMARY:
To find out if adding pembrolizumab to standard of care chemotherapy drugs (cisplatin and gemcitabine) will improve long-term response of intrahepatic cholangiocarcinoma after surgery, compared to treatment with surgery and standard chemotherapy alone.

DETAILED DESCRIPTION:
Primary Objectives and Endpoints:

* To evaluate RFS. RFS will be defined as time from curative-intent surgery to disease recurrence. Median, 9-month, and 12-month RFS rates will be measured.
* To evaluate the rate of major pathologic response. Pathologic response will be assessed both by determining the percentage of the bulk tumor made up of viable cancer cells, with < 10% signifying a major pathologic response, and by evaluating indicators of immune-mediated pathologic response which incorporate elements of tumor necrosis and fibroinflammatory stroma.

Primary Endpoints: RFS rate, major pathologic response rate

Secondary Objectives and Endpoints:

Objectives: To assess safety and other markers of efficacy, including objective response rate (ORR) and overall survival (OS).

Secondary Endpoints:

* To evaluate the safety and efficacy of pembrolizumab in combination with gemcitabine and cisplatin
* Safety profile per CTCAE v5.0, including term, incidence, severity, and duration of AEs
* Objective response rate (ORR) by RECIST 1.1 criteria
* 12- and 24-month overall survival (OS) by RECIST 1.1 criteria
* Median progression free survival (PFS) and median overall survival (OS) according to RECIST v1.1

Exploratory Objectives and Endpoints:

* Correlative studies will be performed to assess the immunologic response to neoadjuvant pembrolizumab with gemcitabine and cisplatin including but not limited to blood and tissue-based biomarkers, gene alterations, immunologic markers and pharmacodynamic markers from study treatment.
* To assess and correlate gut microbiome diversity, composition, structure, and functional characteristics pre- and post-NAT.
* To assess the biliary microbiome diversity, composition and functional characteristics (if bile is able to be collected at the time of surgery), and to compare the biliary microbiome to pre- and post-NAT gut microbiome, as well as to clinicopathologic outcomes.
* To evaluate the effects of pembrolizumab on pharmacodynamic markers: ctDNA, tissue biopsies, and/or blood to assess biomarkers. include, but are not limited to, circulating tumor DNA and exosome analyses, gene expression studies, reverse phase protein arrays (RPPA, and Nanostring and/or RNA-exome to assess mRNA expression.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Provision of signed Informed Consent prior to any screening procedures being performed.
2. Age ≥ 18 years at the time of informed consent.
3. Histologically (or cytologically) confirmed diagnosis of intrahepatic cholangiocarcinoma or adenocarcinoma of suspected biliary origin/ cholangiocarcinoma that is measurable according to RECIST 1.1 criteria.

   a) Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
4. Has high-risk, but resectable, ICC confined to the liver, bile duct, and /or regional lymph nodes. Tumors will be considered high-risk if the high-quality, contrast-enhanced CT and/or MRI +/- positron emission tomography (PET) scan done within 6 weeks of screening show at least one of the following (a-e):

   1. T-stage ≥ Ib (Ib - IIIb)
   2. Solitary lesion > 5 cm
   3. Multifocal tumors or satellite lesions present confined to the same lobe of the liver as the dominant lesion but still technically resectable
   4. Presence of major vascular invasion but still technically resectable
   5. Suspicious or involved regional lymph nodes (N1)
   6. Serum CA 19-9 > 200 U/mL
5. ECOG performance status of 0-1.
6. Adequate hematologic status: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Hemoglobin (Hgb) ≥ 9 g/dL with or without transfusions; Platelets (PLT) ≥ 100 x 109/L without transfusions.
7. Adequate liver function:

   1. ALT and AST ≤2.5 × ULN, or ≤5 × ULN in the presence of liver metastases
   2. Total bilirubin ≤ 1.5 × ULN and < 2 mg/dL i. Note: Patients who have a total bilirubin level > 1.5 x ULN will be allowed if their indirect bilirubin level is ≤ 1.5 x ULN ii. Note: Participants with hyperbilirubinemia due to non-hepatic cause (e.g., hemolysis, hematoma) may be enrolled following discussion and agreement with the principle investigator
   3. International normalized ratio (INR), prothrombin time (PT), Activated partial thromboplastin time (aPTT): ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
8. Adequate renal function: Serum Creatinine ≤ 1.5 x ULN, or calculated creatinine clearance (determined as per Cockcroft-Gault) ≥ 50mL/min at screening.
9. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
10. Participants who are HBsAg positive are eligible if they have received HBV anti-viral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization. Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention. Hepatitis B screening tests are not required unless: known history of HBV infection, or as mandated by local health authority.
11. Participants with a history of HCV infection are eligible if HCV viral load is undetectable at screening. Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization. Hepatitis C screening tests are not required unless: known history of HCV infection, or as mandated by local health authority.
12. Willing and able to participate in the trial and comply with all trial requirements.
13. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational agent may be included after consultation with the medical monitor.
14. The effects of pembrolizumab in combination with gemcitabine and cisplatin on the developing human fetus are unknown. For this reason and because gemcitabine and cisplatin used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

    * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
    * History of hysterectomy or bilateral salpingo-oophorectomy.
    * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
    * History of bilateral tubal ligation or another surgical sterilization procedure.
    * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
    * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study for the duration of study participation, and 4 months after completion of treatment administration.
15. Ability to understand and the willingness to sign a written informed consent document.
16. English and non-English-speaking patients.
17. HIV-infected participants must have well-controlled HIV on ART, defined as:

    * Participants on ART must have a CD4+ T-cell count ≥350 cells/mm3 at the time of screening
    * Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 or the LLOQ (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening
    * It is advised that participants must not have had any AIDS-defining opportunistic infections within the past 12 months.
    * Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (Day 1) and agree to continue ART throughout the study
    * [Include if pembrolizumab or IO/IO combination includes ART that affects CYP] The combination ART regimen must not contain any antiretroviral medications that interact with CYP3A4 inhibitors/inducers/substrates (https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers)

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or antiPDL2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX40, CD137).
2. Has had previous systemic therapy for ICC.
3. Has small cell cancer, neuroendocrine tumors, lymphoma, sarcoma, mixed tumor histology and/or mucinous cystic neoplasm.
4. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.
5. Uncontrolled intercurrent illness including symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia and myocardial infarction (MI) within 3 months of initiation of therapy.
6. Active and uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
7. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
8. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
9. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
11. Known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
12. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
13. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
15. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
16. Has an active infection requiring systemic therapy.
17. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

    Note: Hepatitis B and C screening tests are not required unless:
    * Known history of HBV and HCV infection
    * As mandated by local health authority
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial, as determined by the treating investigator.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
21. Has had an allogenic tissue/solid organ transplant.
22. Cognitive impairment.
23. HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hop Tran Cao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org